CLINICAL TRIAL: NCT06109077
Title: Comparative Effects of Levator Ani Release and Post Isometric Relaxation on Pain, Disability, and Quality of Life Among Patients With Coccydynia
Brief Title: Comparative Effects of Levator Ani Release and Post Isometric Relaxation Among Patients With Coccydynia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0143
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Coccydynia
Keywords: Coccydynia; levator ani; pain; post isometric relaxation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levator ani release (Experimental): Participants will receive levator ani release exercise
  Interventions: Other: Levator ani release
- Post isometric relaxion (Experimental): Participants will receive post isometric relaxion exercise
  Interventions: Other: Post isometric relaxion

INTERVENTIONS:
Other: Levator ani release — Patients will be treated with levator ani release exercises for pain (3 sets with 10 repetitions 3 times per week for 6 weeks).
  Arms: Levator ani release
Other: Post isometric relaxion — Patients will be treated with Post isometric relaxation exercise and hold contractions for 10 seconds over 5 to 12 repetitions, 3 times per week for 6 weeks
  Arms: Post isometric relaxion

SUMMARY:
To compare the effects of levator ani release and post isometric relaxation on pain, disability and quality of life among patients with coccydynia

DETAILED DESCRIPTION:
Coccygodynia, also known as coccalgia, coccygeal neuralgia, or tailbone pain, is the word used to describe the pain symptoms that develop in the coccyx region. The discomfort is typically brought on while the person is sitting down, but it can also start when the person stands up. The majority of instances get well within a few weeks to months, but for certain people, the pain might last longer and have an adverse effect on quality of life. Due to the complexity of coccygeal pain in these people, management can be challenging.

The aim of the study is to compare effects of levator ani release exercises and post isometric in patients with coccydynia. A randomized control trial will be conducted at Jinnah hospital Lahore through convenience sampling technique on 46 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. Group A will be treated with levator ani release exercises and Group B will be treated with post isometric relaxation techniques. Outcome measure will be conducted through pain and disability questionnaire at baseline and after 4 weeks. Data will be analyzed using SPSS software version 21. After assessing normality of data by Shapiro - wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:•

* Both gender
* Age between 20-40 years
* Drivers
* Office workers
* Computer users
* Both gender
* Age between 20-40 years
* Drivers
* Office workers
* Computer users

Exclusion Criteria:

* Neurological disorders,
* Bone deficits,
* Vascular abnormalities,
* Rheumatoid arthritis
* Ankylosing spondylitis
* Fracture
* Tumor

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Pain (NPRS) | 4th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain.
Dallas pain questionnaire (DPQ) | 4th week
  A condition-specific impairment questionnaire as well as pain and satisfaction indicators such self-assessment pain ratings are needed for the evaluation of low back pain (LBP). The 16-item Dallas Pain Questionnaire (DPQ) was created to assess patients' perceptions of the extent to which four parts of their lives are affected by chronic pain. It is simple to comprehend, can be answered in 3 to 5 minutes, and can be scored in under a minute.
Oswestry disability index (ODI) | 4th week
  The ODI comprises of ten items that examine several activities of daily life (such as lifting, walking, and travelling) and measures the limitations of a patient's performance in comparison to that of a fit individual. On a six-point scale, from 0 to 5, each item is scored. By adding together the values of each individual item, dividing that total by the range of potential scores, and multiplying that result by 100, one can approximate the overall ODI score. Higher scores imply greater levels of disability on the scale of 0 to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, Ms, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lirette LS, Chaiban G, Tolba R, Eissa H. Coccydynia: an overview of the anatomy, etiology, and treatment of coccyx pain. Ochsner J. 2014 Spring;14(1):84-7. PMID 24688338
- [Background] Tague RG. Fusion of coccyx to sacrum in humans: prevalence, correlates, and effect on pelvic size, with obstetrical and evolutionary implications. Am J Phys Anthropol. 2011 Jul;145(3):426-37. doi: 10.1002/ajpa.21518. Epub 2011 May 3. PMID 21541925
- [Background] Lawson JO. Pelvic anatomy. I. Pelvic floor muscles. Ann R Coll Surg Engl. 1974 May;54(5):244-52. No abstract available. PMID 4829749
- [Background] Slattengren AH, Nissly T, Blustin J, Bader A, Westfall E. Best uses of osteopathic manipulation. J Fam Pract. 2017 Dec;66(12):743-747. PMID 29202144
- [Background] Enck P, Vodusek DB. Electromyography of pelvic floor muscles. J Electromyogr Kinesiol. 2006 Dec;16(6):568-77. doi: 10.1016/j.jelekin.2006.08.007. Epub 2006 Oct 18. PMID 17055294
- [Background] Mosaad EH, Mohamed AY, Fawzy AA, Mohamed MH. The effect of adding kinesiotaping versus pelvic floor exercise to conventional therapy in the management of post-colonoscopy coccydynia: a single-blind randomized controlled trial. Afr Health Sci. 2023 Mar;23(1):575-583. doi: 10.4314/ahs.v23i1.60. PMID 37545928